CLINICAL TRIAL: NCT02402166
Title: A Phase 2, Open-label, Multicenter, Exploratory Safety, Tolerability, Pharmacokinetic, and Efficacy Study of SPD489 in Preschool Children Aged 4-5 Years With Attention-deficit/Hyperactivity Disorder
Brief Title: Safety, Tolerability, Pharmacokinetic, and Efficacy Study of SPD489 in Preschool Children With Attention-deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD489-211
Record Dates: First submitted 2015-03-19; First posted 2015-03-30 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): There are 4 periods in this study: 1)screening and washout; 2) Dose Optimization; 3) Dose Maintenance; 4) Safety Follow-up. SPD489 will be used to treat all subjects.
  Interventions: Drug: SPD489

INTERVENTIONS:
Drug: SPD489 — All subjects will begin with 5mg of SPD489 daily and will be titrated until optimal dose is reached (5, 10, 15, 20, and 30mg)
  Other Names: Lisdexmfetamine dimesylate

SUMMARY:
The purpose of this study is to gain initial safety, tolerability, pharmacokinetic, and efficacy information on SPD489 in preschool children 4-5 years old who are diagnosed with ADHD. Generating such data will provide data on the use of SPD489 in the preschool ADHD population.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female aged 4-5 years inclusive at the time of consent. Only recruiting male subjects as of December 2015
2. Subject's parent or LAR must provide signature of informed consent, and there must be documentation of assent (if applicable) by the subject in accordance with the ICH GCP Guideline E6 (1996) and applicable regulations, before completing any study-related procedures.
3. Subject and parent/LAR are willing and able to comply with all of the testing and requirements defined in the protocol, including oversight of morning dosing. Specifically, the same parent/LAR should be available daily to dispense the dose of investigational product for the study duration.
4. Subject must meet DSM-IV-TR criteria for a primary diagnosis of ADHD (all subtypes) based on a detailed psychiatric evaluation conducted by a sponsor-approved clinician
5. Subject has an ADHD-RS-IV Preschool Version total score ≥93rd percentile at the Baseline Visit (Visit 0). For boys, this is a score of ≥32. For girls, this is a score of ≥24.
6. Subject has a CGI-S score ≥4 at the Baseline Visit (Visit 0).
7. Subject has a Peabody Picture Vocabulary Test, Fourth Edition standard score of ≥70 at the Screening Visit (Visit -1).
8. Subject has undergone an adequate course of non-pharmacological treatment based on investigator judgment or the subject has a severe enough condition to consider enrollment without undergoing prior non-pharmacological treatment based on investigator judgment.
9. Subject has, in the opinion of the investigator, participated in a structured group activity (e.g., preschool, sports, Sunday school) so as to assess symptoms and impairment in a setting outside the home.
10. Subject has lived with the same parent/LAR for ≥6 months.

Exclusion Criteria:

1. Subject is required to or anticipates the need to take medications that have CNS effects or affect performance, such as sedating antihistamines and decongestant sympathomimetics, or are taking monoamine oxidase inhibitors. Stable use of bronchodilator inhalers is not exclusionary.
2. Subject has taken another investigational product or has taken part in a clinical study within 30 days prior to the Screening Visit (Visit -1).
3. Subject is well controlled on his/her current ADHD medication with acceptable tolerability.
4. Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments conducted in the study or that might increase risk to the subject. Similarly, the subject will be excluded if he or she has any additional condition(s) that, in the investigator's opinion, would prohibit the subject from completing the study or would not be in the best interest of the subject. The additional conditions would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol. Mild, stable asthma is not exclusionary.
5. Subject has failed to fully respond, based on investigator judgment, to a previously administered adequate course of amphetamine therapy.
6. Subject has a documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.
7. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
8. Subject has a blood pressure measurement ≥95th percentile for age, sex, and height at the Screening Visit (Visit -1) or the Baseline Visit (Visit 0).
9. Subject has a known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems placing them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
10. Subject has any clinically significant electrocardiogram at the Screening Visit (Visit -1) or the Baseline Visit (Visit 0) or clinically significant laboratory abnormalities at the Screening Visit (Visit -1) based on investigator judgment.
11. Subject has current abnormal thyroid function, defined as abnormal thyroid stimulating hormone and thyroxine at the Screening Visit (Visit -1). Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
12. Subject has a current diagnosis of adjustment disorder, autism, psychosis, or bipolar disorder.
13. Subject is currently considered at risk for suicide in the opinion of the investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded, based on the assessment of the investigator.
14. Subject has a height ≤5th percentile for age and sex at the Screening Visit (Visit -1).
15. Subject has a weight ≤5th percentile for age and sex at the Screening Visit (Visit -1).
16. Subject has a history of seizures (other than infantile febrile seizures) or a current diagnosis of Tourette's disorder.
17. Subject has a chronic or current tic disorder that is judged by the investigator to be exclusionary.
18. Subject is taking any medication that is excluded.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (6):
- United States (6):
  - AVIDA, Newport Beach, California
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Center For Psychiatry and Behavioral Medicine In, Las Vegas, Nevada
  - Duke Child and Family Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Houston Clinical Trials, LLC, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Childress AC, Findling RL, Wu J, Kollins SH, Wang Y, Martin P, Robertson B. Lisdexamfetamine Dimesylate for Preschool Children with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2020 Apr;30(3):128-136. doi: 10.1089/cap.2019.0117. Epub 2020 Feb 11. PMID 32233956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at seven sites in the United States between 15 Apr 2015 (first participant first visit) and 30 Jun 2016 (last participant last visit).
Pre-assignment Details: A total of 24 participants were enrolled and received at least one dose. Overall 19 participants completed the study.
Groups:
- SPD489: Participants received 5 milligram (mg) capsule of SPD489 orally once daily and titrated up to either 10 mg, 15 mg, 20 mg, or 30 mg until an optimal dose was reached within 8 weeks.
Period: Overall Study
Arm/Group | SPD489
Started | 24
Completed | 19
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all participants who had taken at least 1 dose of investigational product.
Arm/Group | SPD489
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.7 (0.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) at the Specified Dose Level
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An AE was considered treatment-emergent if it had a start date on or after, or had a start date before but increased in severity after the first dose of investigational product.
Time Frame: From start of study treatment up to safety follow-up (Week 9)
Population: Safety analysis set consisted of all participants who had taken at least 1 dose of investigational product. Reporting groups are defined by the dose taken prior to the onset of the TEAE (Treatment Emergent Adverse Event). Number of participants analysed (N) are specific to the reporting group at the specific dose level.
Measure: Count of Participants; unit: Participants
Groups:
- SPD489 5 mg: Participants received 5 mg capsule of SPD489 orally once daily from Week 1 up to Week 8 based on the investigator's assessment of participants' response and tolerability.
- SPD489 10 mg: Participants received 10 mg capsule of SPD489 orally once daily from Week 2 up to Week 8 based on the investigator's assessment of participants' response and tolerability.
- SPD489 15 mg: Participants received 15 mg capsule of SPD489 orally once daily from Week 3 up to Week 8 based on the investigator's assessment of participants' response and tolerability.
- SPD489 20 mg: Participants received 20 mg capsule of SPD489 orally once daily from Week 4 up to Week 8 based on the investigator's assessment of participants' response and tolerability.
- SPD489 30 mg: Participants received 30 mg capsule of SPD489 orally once daily from Week 5 up to Week 8 based on the investigator's assessment of participants' response and tolerability.
- SPD489: Participants received 5 mg capsule of SPD489 orally once daily and titrated up to either 10 mg, 15 mg, 20 mg, or 30 mg until an optimal dose was reached within 8 weeks.
Arm/Group | SPD489 5 mg | SPD489 10 mg | SPD489 15 mg | SPD489 20 mg | SPD489 30 mg | SPD489
Number analyzed (Participants) | 24 | 23 | 18 | 12 | 10 | 24
Participants | 10 | 11 | 7 | 6 | 6 | 19

2. Primary Outcome: Change in Sleep Patterns Assessed by Children's Sleep Habits Questionnaire at Week 8 / End of Treatment (ET)
Description: Children's Sleep Habits Questionnaire is a tool designed to screen the most common sleep problems in children, and consists of 33 items for scoring. The instrument evaluates the child's sleep based on behavior within 8 different subscales: bedtime resistance, sleep-onset delay, sleep duration, sleep anxiety, night walkings, parasomnias, sleep-disordered breathing, and daytime sleepiness. Each item receives a score from 1 (problem occurs rarely) to 3 (problem usually occurs); therefore, a higher score is the worse outcome. Scale ranges are as follows: bedtime resistance: 6 to 18, sleep onset delay: 1 to 3, sleep duration: 3 to 9, sleep anxiety: 4 to 12, night walkings: 3 to 9, parasomnias: 7 to 21, sleep-disordered breathing: 3 to 9, daytime sleepiness: 8 to 24, and total disturbance (items from all scales): 33 to 99.
Time Frame: Baseline, Week 8/ET
Population: Safety analysis set consisted of all participants who had taken at least 1 dose of investigational product. Here number of participant analysed for the each sub-scale is specified for this endpoint.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | SPD489
Number analyzed (Participants) | 24
Units on a Scale
  Baseline : Bedtime resistance | 9.9 (3.58)
  Week 8/ End of Treatment (ET) : Bedtime resistance: number analyzed (Participants) | 22
  Week 8/ End of Treatment (ET) : Bedtime resistance | 9.5 (3.26)
  Baseline : Sleep-onset delay | 1.9 (0.85)
  Week 8/ ET : Sleep-onset delay: number analyzed (Participants) | 22
  Week 8/ ET : Sleep-onset delay | 1.8 (0.92)
  Baseline : Sleep duration | 4.5 (1.56)
  Week 8/ET : Sleep duration: number analyzed (Participants) | 22
  Week 8/ET : Sleep duration | 4.0 (1.27)
  Baseline : Sleep anxiety | 6.6 (2.52)
  Week 8/ET : Sleep anxiety: number analyzed (Participants) | 22
  Week 8/ET : Sleep anxiety | 5.5 (1.79)
  Baseline : Night walkings | 5.0 (2.10)
  Week 8/ET : Night wakings: number analyzed (Participants) | 22
  Week 8/ET : Night wakings | 4.7 (2.00)
  Baseline : Parasomnias | 9.7 (2.03)
  Week 8/ET : Parasomnias: number analyzed (Participants) | 22
  Week 8/ET : Parasomnias | 8.5 (1.57)
  Baseline : Sleep-disordered breathing | 3.3 (0.82)
  Week 8/ET : Sleep-disordered breathing: number analyzed (Participants) | 22
  Week 8/ET : Sleep-disordered breathing | 3.2 (0.66)
  Baseline : Daytime sleepiness | 12.1 (3.43)
  Week 8/ET : Daytime sleepiness: number analyzed (Participants) | 22
  Week 8/ET : Daytime sleepiness | 10.0 (3.51)

3. Primary Outcome: Number of Participants With Suicide Related Behavior Assessed by Columbia-Suicide Severity Rating Scale Questionnaire (C-SSRS)
Description: The C-SSRS is a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behaviour occurred. The interview was initiated with 5 (yes/no) questions, presented in ascending order of severity, about suicidal ideation. The most severe type of ideation was rated for frequency, duration, controllability, deterrents, and reason. If the answer to the first 2 ideation questions was "yes," the clinician asked questions 3-5. Active suicidal ideation included any participant who answered "yes" to questions 2-5. If the answers to ideation questions 1 and 2 were "No," then the clinician proceeded to 5 (yes/no) questions that addressed suicidal behavior, which was categorized as actual attempt, interrupted attempt, aborted attempt, preparatory acts or behaviors, and completed suicide.
Time Frame: Baseline, Week 8/ET
Population: Safety analysis set consisted of all participants who had taken at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | SPD489
Number analyzed (Participants) | 24
Participants | 1

4. Secondary Outcome: Change From Baseline in Attention Deficit/Hyperactivity Disorder Rating Scale (ADHD-RS-IV) Preschool Version Total Score at FoTA (Final on Treatment Assessment)
Description: The ADHD-RS-IV Preschool Version is an 18-item questionnaire that requires the respondent to rate the frequency of occurrence of ADHD symptoms as defined by Diagnostic and Statistical Manual of Mental Disorder, Fourth Edition (DSM-IV-TR) criteria. Each item is scored on a 4-point scale ranging from 0 (never or rarely) to 3 (very often) with total scores ranging from 0-54. The 18 items may be grouped into 2 subscales: hyperactivity/impulsivity (even numbered items 2-18) and inattentiveness (odd numbered items 1-17). Data presented here was analysed at Final on-Treatment Assessment (FoTA).
Time Frame: Baseline, FoTA
Population: Full analysis set consisted of all participants in the safety analysis set who had at least 1 post-dose ADHD-RS-IV Preschool Version total score assessment.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | SPD489
Number analyzed (Participants) | 24
Units on a Scale
  Baseline | 43.6 (5.54)
  FoTA | -26.1 (14.37)

5. Secondary Outcome: Number of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I)
Description: CGI-I was performed to rate the severity of a participant's condition on a 7-point scale (1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; or 7=very much worse). Data presented here was analysed at Final on-Treatment Assessment (FoTA). Improved is defined as a score of "very much improved" or "much improved".
Time Frame: FoTA
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | SPD489
Number analyzed (Participants) | 24
Participants | 20

6. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC 0-last) of SPD489 in Plasma
Description: AUC 0-last is the area under the concentration-time curve from time zero to the time of the last quantifiable concentration of SPD489 in plasma. Pharmacokinetic (PK) parameters were compared against the study NRP104-201 (NCT00557011) to observe and compare the effects of SPD489.
Time Frame: Visit 7 [Dose Maintenance Phase] at pre-dose, and 1, 2, 3, 4, 6, and 8 h post-dose
Population: The PK set consisted all participants in the safety analysis set for whom the primary PK data were considered sufficient and interpretable. PK assessments were performed only during the Dose Maintenance Period (2 weeks) for SPD 489 10, 15 and 30 mg reporting groups.
Measure: Mean (Standard Deviation); unit: hour*nanogram/millilitre(h*ng/mL)
Arm/Group | SPD489 10 mg | SPD489 15 mg | SPD489 30 mg
Number analyzed (Participants) | 1 | 2 | 5
hour*nanogram/millilitre(h*ng/mL) | 9.8 (NA) — Due to insufficient number of subject (N=1), standard deviation value was not calculated. | 15.7 (4.1) | 59.5 (22.0)

ADVERSE EVENTS:
Time Frame: From Start of Treatment up to Safety Follow up (Week 9)
Groups:
- SPD489 5mg: Participants received 5 mg capsule of SPD489 orally once daily from Week 1 up to Week 8 based on the investigator's assessment of participants' response and tolerability.
- SPD489 10mg: Participants received 10 mg capsule of SPD489 orally once daily from Week 2 up to Week 8 based on the investigator's assessment of participants' response and tolerability.
- SPD489 15mg: Participants received 15 mg capsule of SPD489 orally once daily from Week 3 up to Week 8 based on the investigator's assessment of participants' response and tolerability.
- SPD489 20mg: Participants received 20 mg capsule of SPD489 orally once daily from Week 4 up to Week 8 based on the investigator's assessment of participants' response and tolerability.
- SPD489 30mg: Participants received 30 mg capsule of SPD489 orally once daily from Week 5 up to Week 8 based on the investigator's assessment of participants' response and tolerability.
Arm/Group | SPD489 5mg | SPD489 10mg | SPD489 15mg | SPD489 20mg | SPD489 30mg | SPD489
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/18 | 0/12 | 0/10 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/18 | 0/12 | 0/10 | 0/24
Other Adverse Events (participants affected / at risk) | 6/24 | 7/23 | 7/18 | 6/12 | 6/10 | 15/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD489 5mg (N=24) | SPD489 10mg (N=23) | SPD489 15mg (N=18) | SPD489 20mg (N=12) | SPD489 30mg (N=10) | SPD489 (N=24)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 8 (8)
Affect lability (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 4 (6)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Middle insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.